CLINICAL TRIAL: NCT02466425
Title: A Phase 3, Randomized, Double-blind, Multi-center, Placebo Controlled, Dose-Optimization, Safety and Efficacy Study of SHP465 in Children and Adolescents Aged 6-17 Years With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy Study of SHP465 in Children and Adolescents Aged 6-17 Years With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHP465-305
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHP465 (Experimental): Subjects will receive SHP465 (12.5mg and 25mg capsules) or matching placebo. Subjects will take 1 capsule daily throughout the study at approximately 7:00am (+/- 2 hours)
  Interventions: Drug: SHP465
- Placebo (Placebo Comparator): Subjects will receive SHP465 (12.5mg and 25mg capsules) or matching placebo. Subjects will take 1 capsule daily throughout the study at approximately 7:00am (+/- 2 hours)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHP465 — 12.5mg and 25mg capsules (one capsule daily)
  Arms: SHP465
Drug: Placebo — Matching placebo capsule that appear identical in size, weight, shape, color
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the efficacy and safety of SHP465 in the treatment of ADHD in children and adolescents (aged 6-17 years). The primary objective of this study is to evaluate the efficacy of SHP465 administered as a daily morning dose compared to placebo in the treatment of children and adolescents (6-17 years of age inclusive) diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 6-17 years of age, inclusive, at the time of consent.
2. Subject's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions in accordance with the ICH GCP Guideline E6 (1996) and applicable regulations before completing any study-related procedures.
3. Subject and parent/LAR are willing and able to comply with all of the testing and requirements defined in the protocol, including oversight of morning dosing. Specifically, the parent/LAR must be available at approximately 7:00AM (±2 hours) to dispense the dose of investigational product for the study duration.
4. Subject, who is a female and of child-bearing potential, must not have a positive serum beta human chorionic gonadotropin pregnancy test at the Screening Visit (Visit 1) and must have a negative urine pregnancy test at the Baseline Visit (Visit 2) and agree to comply with any applicable contraceptive requirements of the protocol.
5. Subject must have a satisfactory medical assessment with no clinically significant or relevant abnormalities.
6. Subject meets DSM-IV-TR criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation.
7. Subject has an ADHD-RS-IV Total Score >28 at the Baseline Visit (Visit 2).
8. Subject is functioning at an age-appropriate level intellectually, as determined by the study Investigator.
9. Subject is currently not on ADHD therapy, or is not completely satisfied with any aspect of their current ADHD therapy.
10. Subject is able to swallow a capsule whole.

Exclusion Criteria:

1. Subject has a current, controlled (with medications prohibited in this study) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any significant comorbid Axis II disorder or significant Axis I disorder (such as post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, depressive or anxiety disorder) or other symptomatic manifestations that, in the opinion of the examining clinician, will contraindicate treatment with SHP465 or confound efficacy or safety assessments. Comorbid psychiatric diagnoses will be established with the Screening Visit (Visit 1) interview of the K-SADS-PL and additional modules if warranted by the results of the initial interview. Subjects may continue participation in a behavioral modification program during the study as long as they have been participating in the program for at least 1 month at the time of the Baseline Visit (Visit 2).
2. Subject meets DSM-IV-TR diagnosis of conduct disorder. Oppositional defiant disorder is not exclusionary.
3. Subject is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.
4. Subject is underweight based on Centers for Disease Control and Prevention body mass index (BMI)-for-age sex-specific values at the Screening Visit (Visit 1). Underweight is defined as a BMI <3rd percentile
5. Subject is significantly overweight based on Centers for Disease Control and Prevention BMI-for-age sex specific values at the Screening Visit (Visit 1). Significantly overweight is defined as a BMI >97th percentile for this study
6. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that, in the Investigator's opinion, would prohibit the subject from completing the study or would not be in the best interest of the subject. The additional conditions would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
7. Subject has a history of seizure (other than infantile febrile seizures), a chronic or current tic disorder, or a current diagnosis of Tourette's Disorder. Subject has a history of tics that are judged by the Investigator to be exclusionary.
8. Subject's blood pressure measurements exceed the 90th percentile for age, sex, and height (based on the Blood Pressure Levels by Age and Height Percentile [for boys and girls]) at the Screening Visit (Visit 1) and the Baseline Visit (Visit 2)
9. Subject has a known history of hypertension
10. Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place him/her at increased vulnerability to the sympathomimetic effects of a stimulant medication.
11. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
12. Subject has any clinically significant ECG or clinically significant laboratory abnormality at the Screening Visit (Visit 1).
13. Subject has current abnormal thyroid function, defined as abnormal thyroid stimulating hormone and thyroxine at the Screening Visit (Visit 1). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
14. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
15. Subject has failed to respond, based on Investigator judgment, to an adequate course(s) (dose and duration) of amphetamine therapy
16. Subject has a history of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR criteria. Subjects with a lifetime history of amphetamine, cocaine, or other stimulant abuse and/or dependence will be excluded.
17. Subject has a positive urine drug result at the Screening Visit (Visit 1) (with the exception of subject's current stimulant therapy, if any) or the Baseline Visit (Visit 2), if repeated unless the Investigator can verify that the positive result at the Screening Visit (Visit 1) is attributed to medication that has been prescribed to the subject and will be discontinued prior to the Baseline Visit (Visit 2). A positive result at the Screening Visit (Visit 1) attributed to a prescribed medication requires a re-test and a negative result at the Baseline Visit (Visit 2) to confirm subject eligibility.
18. Subject has taken another investigational product or has taken part in a clinical study within 30 days prior to the Screening Visit (Visit 1).
19. Subject has previously completed, discontinued, or was withdrawn from this study.
20. Subject is taking any medication that is excluded or has not been appropriately washed out according to the protocol requirements.
21. Subject is required to take or anticipates the need to take medications that have central nervous system effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
22. Subject is female and is pregnant or lactating

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2016-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (36):
- United States (36):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Nrc Research Institute, Orange, California
  - Pcsd Feighner Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - McB Clinical Research Centers, Colorado Springs, Colorado
  - Florida Clinical Research Center, Llc, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, Llc, South Miami, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group Inc, Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - Rochester Center For Behavioral Medicine, Rochester Hills, Michigan
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Center For Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Midwest Clinical Research Center, Dayton, Ohio
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Oregon Center For Clinical Investigations, Inc, Salem, Oregon
  - Omega Medical Research, Warwick, Rhode Island
  - Rainbow Research, Barnwell, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solution, Inc, Memphis, Tennessee
  - Futuresearch Trials of Dallas, Lp, Dallas, Texas
  - Bayou City Research, Houston, Texas
  - Red Oak Psychiatry Associates, Pa, Houston, Texas
  - Houston Clinical Trials, Llc, Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Research Across America, Plano, Texas
  - Eastside Therapeutic Resource, Kirkland, Washington

REFERENCES:
- [Result] Brams M, Childress AC, Greenbaum M, Yu M, Yan B, Jaffee M, Robertson B. SHP465 Mixed Amphetamine Salts in the Treatment of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents: Results of a Randomized, Double-Blind Placebo-Controlled Study. J Child Adolesc Psychopharmacol. 2018 Feb;28(1):19-28. doi: 10.1089/cap.2017.0053. Epub 2017 Aug 17. PMID 28816509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 36 sites in the United States between 18 June 2015 and 16 February 2016.
Pre-assignment Details: A total of 338 participants were screened and 264 participants were enrolled in the study.
Groups:
- Placebo: Participants received placebo matched to SHP465 capsule orally once daily for 4 weeks.
- SHP465: Participants received SHP465 capsule (12.5 milligram [mg] during dose optimization and 25 mg during the dose maintenance phase) orally once daily for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | SHP465
Started | 132 | 132
Treated | 131 | 132
Completed | 118 | 116
Not Completed | 14 | 16
Not completed — Adverse Event | 3 | 11
Not completed — Lack of Efficacy | 4 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 1 | 3
Not completed — Withdrawal by Parent/Guardian | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants in the randomized set (participants who signed informed consent for whom a randomization number had been assigned) who had taken at least 1 dose of investigational product.
Groups:
- SHP465: Participants received SHP465 capsule (12.5 mg during dose optimization and 25 mg during the dose maintenance phase) orally once daily for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | SHP465 | Total
Number analyzed (Participants) | 131 | 132 | 263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.5 (3.24) | 12.4 (3.25) | 12.5 (3.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 46 | 100
  Male | 77 | 86 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention-Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Total Score at Visit 6 (Week 4)
Description: The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD based on diagnostic and statistical manual of mental disorders, fourth edition - text revision (DSM-IV-TR) criteria. Each item is scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items may be grouped into 2 subscales: hyperactivity/impulsivity (even-numbered items 2-18) and inattentiveness (odd-numbered items 1-17). Higher score = more severe symptoms.
Time Frame: Baseline, Visit 6 (Week 4)
Population: Full-analysis set (FAS) consisted of the safety set who had at least 1 post-dose ADHD-RS-IV total score assessment. FAS with number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 129 | 128
Units on a scale
  Baseline | 40.0 (6.96) | 39.0 (6.95)
  Change at Visit 6 (Week 4): number analyzed (Participants) | 117 | 113
  Change at Visit 6 (Week 4) | -11.7 (13.37) | -21.5 (11.53)
Statistical Analysis 1: Comparison: Placebo vs SHP465; Test type: Superiority or Other; p < 0.001, Mixed-effects model for repeated measure; LS Mean difference = -9.9, 95% CI 2-sided [-13.0 to -6.8], Standard Error of Mean 1.59 — Between treatment groups

2. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Visit 6 (Week 4)
Description: CGI-I was performed to rate the severity of a participant's condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Visit 6 (Week 4)
Population: FAS with number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | SHP465
Number analyzed (Participants) | 117 | 112
Units on a scale | 2.9 (1.20) | 2.1 (1.13)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to safety follow-up assessment (35 days)
Groups:
- SHP465: Participants received SHP465 capsule (12.5 mg during dose optimization and 25 mg during dose maintenance phase) orally once daily for 4 weeks.
Arm/Group | Placebo | SHP465
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/132
Other Adverse Events (participants affected / at risk) | 26/131 | 67/132
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=131) | SHP465 (N=132)
Nausea (Gastrointestinal disorders) | 4 (5) | 9 (10)
Weight decreased (Investigations) | 1 (1) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 40 (44)
Headache (Nervous system disorders) | 14 (18) | 16 (18)
Insomnia (Psychiatric disorders) | 2 (2) | 15 (17)
Irritability (Psychiatric disorders) | 2 (2) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.